CLINICAL TRIAL: NCT06797531
Title: Real-world Evidence Non-Interventional proSpective Study of kisqaLi (Ribociclib) Effectiveness and safEty in Patients With HR+/HER2- Early Breast Cancer in Saudi Arabia
Brief Title: RWE Non-Interventional Prospective Study of Ribociclib Effectiveness and Safety in Patients With HR+/HER2- Early Breast Cancer in Saudi Arabia
Acronym: NISLEESA
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLEE011ASA01
Record Dates: First submitted 2025-01-21; First posted 2025-01-28 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: HR+/HER2- Early Breast Cancer
Keywords: Early breast cancer; Saudi Arabia; Ribociclib; Effectiveness; Safety; Real world evidence; RWE; Observational study
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Ribocliclib: HR+/HER2- early breast cancer patients who have been newly receiving ribociclib for up to 6 months prior to enrollment
  Interventions: Drug: ribociclib

INTERVENTIONS:
Drug: ribociclib — This is an observational study. There is no treatment allocation. The decision to initiate ribociclib will be based solely on clinical judgement.

SUMMARY:
This is a non-interventional, prospective, single-arm, observational study describing the real-world effectiveness, safety, and PRO and HCRU data of ribociclib combined with adjuvant ET under conditions of routine clinical practice in HR+/HER2- EBC in premenopausal, perimenopausal and postmenopausal women, or men in Saudi Arabia.

DETAILED DESCRIPTION:
This is a non-interventional, prospective, single-arm, observational study describing the real-world effectiveness, safety, and PRO and HCRU data of ribociclib combined with adjuvant ET under conditions of routine clinical practice in HR+/HER2- EBC in premenopausal, perimenopausal, and postmenopausal women or men in Saudi Arabia.

The study aims to recruit 177 patients who have been newly receiving ribociclib for up to 6 months prior to enrollment date, as per the locally approved label to which the physician has made an independent decision to prescribe ribociclib. Patients will be enrolled over a recruitment window of 9 months and will be followed up for 36 months to assess the study outcomes. It is planned to capture data at the following timepoints (+/- 1 month): Baseline, 3, 6, 12, 24, and 36 months. This is in line with the frequency of routine follow-up visits, per standard of care.

Data will be collected from patients' electronic medical records in the selected sites. The planned number of sites is 6, to be selected based on feasibility reports, considering the patient pool and research capabilities.

Participating sites' investigators will review all the available clinical files of patients whose ribociclib treatment decision has been made by their treating physician and will invite those who fulfill the eligibility criteria to participate in the study. Data will be entered into an electronic case report form (eCRF). All patients' data will remain anonymized, fulfilling the requirements of data protection. Data collected will include information on previous treatments received, disease history, and current treatment patterns and outcomes.

Participation in the study is not intended to change the routine treatment patients receive as determined by their treating physicians; all therapeutic decisions, as well as the type and timing of disease monitoring, will be at the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated Patient Informed Consent Form (PICF) obtained.
2. The patient is ≥ 18 years-old at the time of PICF signature.
3. Male or female patients with estrogen-receptor-positive and/or progesterone-receptor-positive BC.
4. Male or female patients with HER2- BC.
5. Patients who are currently receiving ribociclib in combination with adjuvant ET as per approved local label for up to 6 months prior the enrollment date.
6. Male or female patients with American Joint Committee on Cancer (AJCC) Anatomic Stage Group IIA(subset) /IIB or Anatomic Stage Group III EBC.
7. Female patients with known menopausal status (at the time of PICF signature or initiation of adjuvant ET, whichever occurs earlier), or male.

Exclusion Criteria:

1. Ribociclib-based treatment regimen beyond adjuvant therapy for EBC.
2. Patients are currently participating in any other clinical trials.
3. Patients who previously received any other CDK4/6 inhibitor.
4. Patients who refused to sign informed consent.
5. According to the investigator's opinion, the patient is an unlikely candidate to provide an accurate medical history and/or to obtain long-term follow-up information for any reason.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HR+/HER2- early breast cancer in premenopausal, perimenopausal, and postmenopausal women or men in Saudi Arabia.
Sampling Method: Non-Probability Sample
Enrollment: 177 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Invasive Breast Cancer-Free Survival (iBCFS) | 36 months
  iBCFS, defined as the time from the date of first dose to the date of the first event of invasive ipsilateral breast tumor recurrence, local/regional invasive recurrence, distant recurrence, death (any cause), or invasive contralateral BC.
  iBCFS will be assessed using STEEP Version 2.0 criteria (Standardized Definitions for Efficacy Endpoints in Adjuvant BC Clinical Trials), as assessed by the investigator, in patients with HR+/HER2- Anatomic Stage Group IIA(subset)/IIB/III EBC.

SECONDARY OUTCOMES:
Invasive disease free survival (iDFS) | Up to 36 months
  iDFS is a composite endpoint that contains invasive Ipsilateral Breast Tumor Recurrence (IBTR), loco-regional invasive recurrence, distant recurrence, death from BC, death from non-BC cause, death from unknown cause, invasive contralateral BC and second primary invasive cancer (non-breast) in patients with HR+/HER2- Anatomic Stage Group IIA(subset)/IIB//III EBC.
Distant disease free survival (DDFS) | Up to 36 months
  DDFS defined as distant recurrence, death from BC, death from non-BC cause, death from unknown cause and second primary invasive cancer (non-breast) in patients with HR+/HER2- Anatomic Stage Group IIA(subset)/IIB/III EBC.
Frequency and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | 36 months
  Frequency and severity of AEs and SAEs including laboratory findings, AST/ALT elevations and ECG abnormalities qualifying and reported as AEs.
Change from baseline in the physical functioning sub-scale score and global health status/QoL scale score as assessed by EORTC QLQ-C30 | 36 months
  European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire (EORTC QLQ-C30) incorporates nine multi-item scales: five functional scales (Physical, Role, Cognitive, Emotional and Social Functioning); three symptom scales (Fatigue, Pain and Nausea/Vomiting); and a Global Health Status/QoL scale. Six single item scales are also included (Dyspnoea, Insomnia, Appetite Loss, Constipation, Diarrhoea and Financial Difficulties). All of the scales range in score from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning whereas a high score for a symptom scale or item represents a high level of symptomatology or problems.
Demographics - Age | Baseline
  Age at baseline (years)
Demographics - Gender, race, region | Baseline
  Number of participants per gender, race and region
Clinical characteristics - menopausal status | Baseline up to 36 months
  Assessment of menopausal status
Clinical characteristics - anatomical stage | Baseline up to 36 months
  Assessment of anatomical stage (IIa/IIb/III) according to American Joint Committee on Cancer (AJCC)
Clinical characteristics - pre-index chemotherapy and concomitant medication | Baseline up to 36 months
  Assessment of pre-index chemotherapy and concomitant medications
Clinical characteristics - medical history | Baseline up to 36 months
  Assessment of medical history

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Riyadh, Saudi Arabia